CLINICAL TRIAL: NCT06921421
Title: Assessment Of Burn Severity and Extent Spatial Frequency Domain Imaging (SFDI): An Observational Pilot Study
Brief Title: Assessment Of Burn Severity and Extent Spatial Frequency Domain Imaging
Status: Not yet recruiting | Type: Observational
Sponsor: The Metis Foundation (Other)
Collaborators: The United States Institute of Surgical Research (Unknown); Modulated Imaging Inc. (Industry)
Responsible Party: Principal Investigator, Rodney Chan, Principal Investigator, The Metis Foundation
Other Study IDs: H-25-017; MTEC-22-08-BDA-007 (Other Grant/Funding Number: Medical Technology Enterprise Consortium)
Record Dates: First submitted 2025-03-07; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Burn; Burn Injury
Keywords: SFDI; Spatial Frequency Domain Imaging; Burn depth; Burn injury assessment
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Spatial Frequency Domain Imaging — Spatial Frequency Domain Imaging captures at specific timepoints.

SUMMARY:
The goal of this pilot clinical study is to evaluate the feasibility of collecting Spatial Frequency Domain Imaging (SFDI) data in patients with circulatory compromise due to thermal burns using the FDA-cleared Clarifi Imaging System and the next generation handheld m-Clarifi. Accurate assessment of burn depth and assessment at the point of care is an essential input for clinicians to plan proper treatment and management. SFDI has been shown to be a promising method to evaluate burn depth and extent within 24 hours in pre-clinical studies. The two feasibility goals of this study are as follows: 1) Do the values obtained with a commercial SFDI system provide utility in assessing burn depth in a clinical setting? And 2) Do Clarifi and m-Clarifi provide equivalent data when assessing subjects with burn injuries (biomarker imaging values, clinical workflow).

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. Thermal burns of any depth (superficial, deep partial thickness, or full thickness).

Exclusion Criteria:

1. Patients less than 18 years of age
2. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving care at the US Army Institute of Surgical Research (USAISR) Burn Center with thermal burn injuries will be considered for enrollment into this study
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean SFDI Scattering Parameter (mm-¹) at Burn Injury Sites Using Clarifi and m-Clarifi Imaging Systems | From enrollment to 21 days
  This outcome will report the mean value of the scattering coefficient (μs'), a quantitative SFDI-derived biomarker that correlates with burn depth, measured at specified time points (Day 0, 3, 7, 14, and 21) using the Clarifi and m-Clarifi imaging systems. Higher scattering values are associated with deeper tissue damage.

SECONDARY OUTCOMES:
Correlation Between SFDI Scattering Parameter and Clinician-Determined Burn Depth | From enrollment to 21 days
  This outcome evaluates the statistical correlation between SFDI scattering values and the burn depth classifications made by clinicians based on visual assessment and standard clinical criteria (e.g., superficial partial, deep partial, full thickness).

OTHER OUTCOMES:
Agreement Between Clarifi and m-Clarifi Devices in Measuring SFDI Scattering Parameter | From enrollment to 21 days
  This outcome assesses the agreement between SFDI scattering measurements obtained from the Clarifi (FDA-cleared) and m-Clarifi (handheld prototype) devices at the same anatomical burn sites. Agreement will be quantified using Bland-Altman analysis and intraclass correlation coefficients (ICCs).

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Chan, MD, Principal Investigator — The Metis Foundation
Locations (1):
- The United States Army Institute of Surgical Resarch, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided